CLINICAL TRIAL: NCT06492304
Title: A Phase 1/2 Dose Evaluation and Cohort Expansion Study of the Safety and Efficacy of Anti-CD70 Allogeneic CRISPR-Cas9-Engineered T Cells (CTX131) in Adult Subjects With Relapsed/Refractory Hematologic Malignancies
Brief Title: A Safety and Efficacy Study Evaluating CTX131 in Adult Subjects With Relapsed/Refractory Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-008
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: T Cell Lymphoma; B Cell Lymphoma; Acute Myeloid Leukemia
Keywords: CAR T; B Cell Lymphoma; T Cell Lymphoma; Allogeneic; Leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, B-Cell; Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CTX131 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy
  Interventions: Biological: CTX131

INTERVENTIONS:
Biological: CTX131 — CTX131 (CD70-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components

SUMMARY:
This is an open label, multicenter, phase 1/2 dose evaluation and cohort expansion study evaluating the safety and efficacy of CTX131 in subjects with Relapsed/Refractory Hematologic Malignancies

DETAILED DESCRIPTION:
The study may enroll up to 290 subjects in total. CTX131 is a CD70-directed chimeric antigen receptor (CAR) T cell immunotherapy comprised of allogeneic T cells prepared for the treatment of relapsed/refractory hematological malignancies. The cells are from healthy adult volunteer donors that are genetically modified ex vivo using CRISPR-Cas9 (clustered regularly interspaced short palindromic repeats/ CRISPR-associated protein 9) gene editing components (single guide RNA and Cas9 nuclease)

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (ECOG status of 2 will be permitted for subjects with AML)
3. Diagnosed with r/r T Cell Lymphoma (TCL), B Cell Lymphoma (BCL), or Acute Myeloid Leukemia (AML) T cell lymphoma, including Stage ≥IIB Mycosis fungoides (MF)/ Sézary syndrome (SS) after at least 2 prior systemic therapies Peripheral T cell lymphoma (PTCL) after at least 1 prior line of therapy (PTCL-note otherwise specified (NOS), PTCL-T follicular helper (TFH), Angioimmunoblastic T cell lymphoma (AITL), Adult T cell leukemia/lymphoma (ATLL) of leukemic, lymphomatous, and chronic unfavorable subtypes), (ALK)- ALCL after at least 1 prior line of therapy, ALK+ Anaplastic large cell lymphoma (ALCL) after at least 2 prior lines of therapy

   B cell lymphoma, including Diffuse large B cell lymphoma (DLBCL)-NOS, transformed marginal zone lymphoma(MZL), transformed FL, high-grade BCL with MYC and BCL2 and/or BCL6 rearrangements, Follicular lymphoma (FL) grade 3b, after at least 2 prior lines of therapy including an anti- CD20 monoclonal antibody and an anthracycline containing regimen Mantle cell lymphoma (MCL) after up to 5 prior lines of therapy which must include an anthracycline- or bendamustine-containing regimen, an anti- CD20 monoclonal antibody, and a BTK inhibitor

   Acute myeloid leukemia or AML/MDS per ELN criteria 2022 after at least 1 prior line of AML therapy. APL, BCR-ABL positive leukemia, and AML secondary to prior therapy or history of genetic syndrome associated with BM failure are excluded.
4. Adequate renal, liver, cardiac and pulmonary organ function
5. Females of childbearing potential and male subjects must agree to use an acceptable, highly effective method of contraception (as specified in the protocol) from enrollment through at least 12 months after last CTX131 infusion

Exclusion Criteria:

1. Prior treatment with anti-CD70 targeting agents
2. Active CNS manifestation of underlying disease
3. History or presence of clinically relevant CNS pathology such as seizure, stroke, severe brain injury, cerebellar disease, myelopathy, history of posterior reversible encephalopathy syndrome with prior therapy, or another condition that in opinion of investigator may increase CAR T-related toxicities
4. Uncontrolled bacterial, viral, or fungal infection
5. Positive for HIV, or active hepatitis B virus or hepatitis C virus infection.
6. Concurrent systemic treatment with an anticancer biologic (e.g., monoclonal antibody) within 30 days prior to CTX131 infusion or with a non-biological anticancer drug within 14 days prior to CTX131 infusion. Mogamulizumab treatment is prohibited 50 days prior to CTX131 infusion.
7. Diagnosis with another invasive malignancy in the last 5 years with the exception of non- melanoma skin cancer and malignancies deemed by the investigator and medical monitor to be of low likelihood for recurrence
8. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
9. Prior solid organ or allogeneic BM transplantation, except for AML cohorts if at least 3 months since allogeneic HSCT, not receiving immunosuppressive therapy or donor lymphocyte infusion post SCT in the 2 weeks prior to lymphodepletion, and have no clinically active GvHD
10. Treatment with CD19-targeting CAR-T within 6 months prior to CTX131 infusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Part A (dose escalation) and Part B (dose optimization in selected disease types): | From CTX131 infusion up to 28 days post-infusion
  For all cohorts: Incidence of Adverse events defined as dose-limiting toxicities
Objective Response rate (ORR) | From CTX131 infusion up to 60 months post-infusion
  Phase 2 (expansion of selected Phase 1 disease types)
Composite Complete Remission (CRc) | From CTX131 infusion up to 60 months post-infusion
  Phase 2 (expansion of selected Phase 1 disease types)

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Keegan, MD, PhD, Study Director — CRISPR Therapeutics
Locations (7):
- United States (6):
  - Research Site 6, Phoenix, Arizona
  - Research Site 5, Stanford, California
  - Research Site 3, Boston, Massachusetts
  - Research Site 4, New York, New York
  - Research Site 2, The Bronx, New York
  - Research Site 1, Houston, Texas
- Research Site 7, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No